CLINICAL TRIAL: NCT01104077
Title: Family and Personal History of Pancreatic and Other Malignancies in Patients With Intraductal Papillary Mucinous Neoplasms
Brief Title: Family and Personal History of Malignancy in Intraductal Papillary Mucinous Neoplasm (IPMN)
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAD6106
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Pancreatic Cancer; Neoplasm
Keywords: Pancreatic Cancer; Family History; Pre-cancerous lesion; Intraductal Papillary Mucinous Neoplasm (IPMN); Intraductal Papillary Mucinous Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a retrospective observational study to determine the proportion of patients with a family history of pancreatic cancer and other malignancies among patients who have intraductal papillary mucinous neoplasm (IPMN).

The investigators will be reviewing the demographic, clinical, radiologic, pathologic, and follow-up information from the Pancres Center database. The investigators will also conduct a chart review to collect information recorded by clinicians on each subject's family history of malignancy and personal history of malignancy. Results of this database and chart review will be incorporated into a datasheet in which all patient identifiers have been removed.

The primary outcome will be the percentage of IPMN patients with at least one first-degree relative with pancreatic cancer or IPMN, or at least two first or second degree relatives with pancreatic cancer, IPMN, or malignancies related to pancreatic cancer syndromes, including colorectal, gastric, breast, ovarian, and melanoma neoplasms. Secondary outcomes will be the relative risk of IPMN subtypes of higher malignant potential (main duct or mixed type location), more advanced histology (carcinoma in situ or invasive carcinoma), and recurrence following surgical resection amongst subjects with a family history.

DETAILED DESCRIPTION:
Intraductal papillary mucinous neoplasm (IPMN) is a cyst-like cancer of the pancreas that is increasingly being identified in medical practice, including during the screening of individuals at high risk of pancreatic cancer. It has been established that 10 to 20% of pancreatic cancers are familial. In comparison, there has been little research into the importance of genetic risk in IPMN incidence. The investigators will perform a retrospective chart review of patients with IPMN who were evaluated for surgical intervention at our tertiary referral center. The investigators are interested in determining the proportion of IPMN patients with a family history of pancreatic and other cancers. In addition, the investigators will assess if familial cancer risk is associated with increased risk for malignant IPMN and recurrence, relative to those patients without an inherited predisposition.

ELIGIBILITY:
Inclusion Criteria:

* Tissue-confirmed diagnosis of intraductal papillary mucinous neoplasm or imaging suspicious for IPMN
* Seen in consultation for IPMN at Columbia-Presbyterian Medical Center between 2002 and 2008

Exclusion Criteria:

* Not meeting the inclusion criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Columbia University Medical Center's Pancreas Center who have been diagnosed with intraductal papillary mucinous neoplasm, a cystic neoplasm of the pancreatic duct that has malignant potential.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2008-11-17 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Percentage of IPMN patients with relatives with pancreatic cancer or IPMN | 20 years
  Extent of Family History: The primary outcome will be the percentage of IPMN patients with at least one first-degree relative with pancreatic cancer or IPMN, or at least two first or second degree relatives with pancreatic cancer, IPMN, or malignancies related to pancreatic cancer syndromes, including colorectal, gastric, breast, ovarian, and melanoma neoplasms.

SECONDARY OUTCOMES:
Percentage of IPMN patients exhibiting higher malignant potential or recurrence following surgical resection | 20 years
  Characteristics of IPMN patients with Family History: Secondary outcomes will be the relative risk of IPMN subtypes of higher malignant potential (main duct or mixed type location), more advanced histology (carcinoma in situ or invasive carcinoma), and recurrence following surgical resection amongst subjects with a family history.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K Chung, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No